CLINICAL TRIAL: NCT05933226
Title: A Stepped Care, Peer-Delivered Intervention to Improve ART Adherence and SUD in Primary Care
Brief Title: Project Khanya: Peer-Delivered Intervention to Improve HIV Medication Adherence and Substance Use in South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Cape Town (Other); National Institute on Drug Abuse (NIDA) (NIH); Weill Medical College of Cornell University (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 077/2022; R01DA056102 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Human Immunodeficiency Virus; Alcohol-Related Disorders; Drug Use; Substance Use
Keywords: Immunologic Deficiency Syndrome; Substance Use; Acquired Immunodeficiency Syndrome; Immune system diseases; behavioral symptoms; RNA Virus Infections; HIV Infections; Alcohol Use; Drug Use; Treatment Adherence and Compliance; Delivery and Health Care; Task Sharing; Mental Health; Global Health; South Africa; Cost Effectiveness; Implementation Science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol-Related Disorders; Substance-Related Disorders; Immunologic Deficiency Syndromes; Immune System Diseases; Behavioral Symptoms; RNA Virus Infections; HIV Infections; Alcohol Drinking; Treatment Adherence and Compliance; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Khanya (Experimental): Khanya is a peer-delivered, behavioral intervention to improve HIV medication adherence and reduce problematic SUD symptoms. Khanya is delivered as a stepped-care package in which the least resource-intensive part of the intervention (i.e., Life-Steps, a single session problem solving intervention for HIV medication adherence) will be delivered first. Only individuals randomized to the Khanya intervention who are still struggling with HIV medication adherence after the first session will be stepped up to receive the more comprehensive, resource-intensive part of the intervention (i.e., six additional sessions of the intervention). Khanya Step 2 includes evidence-based treatment components to improve ART adherence and SUD, including motivational interviewing, behavioral activation, and mindfulness-based relapse prevention strategies, which have previously been piloted in this community.
  Interventions: Behavioral: Khanya
- Enhanced Standard of Care (ESOC) (No Intervention): Enhanced Standard of Care (ESOC) includes the local standard of care, which is referral to a free local outpatient substance use treatment program, enhanced with facilitated referrals. To enhance the standard of care, study staff will provide participants with a detailed description of the program's referral process and offer to help the participant set up an intake at the program. Additionally, the team will follow up on the referral.

INTERVENTIONS:
Behavioral: Khanya — "Khanya" is a peer-delivered, behavioral intervention to improve HIV medication adherence and reduce problematic SUD symptoms. Participants will either receive Khanya Step 1 or if they continue to struggle with ART adherence, they will be stepped up to the more intensive intervention, Khanya Step 2.
  Arms: Khanya

SUMMARY:
The purpose of this study is to evaluate a stepped care behavioral intervention for HIV medication adherence and substance use ("Khanya") integrated into an HIV primary care setting in South Africa. The intervention is specifically designed to be implemented by non-specialist counselors with lived substance use experience (i.e., peers), using a task sharing, stepped care model in local primary care clinics. The Khanya stepped care package will be compared to usual care, enhanced with referral to a local outpatient substance use treatment program (Enhanced Standard of Care - ESOC) over 12 months.

DETAILED DESCRIPTION:
South Africa is home the highest number of people living with HIV in the world and has a high burden of substance use disorder (SUD). Globally, a SUD treatment gap exists, particularly in low and middle-income countries (LMICs), such as South Africa, where only 1-4% of individuals receive minimally adequate treatment. Workforce shortages are also severe in LMICS, and countries such as South Africa have responded to this through the implementation of task sharing models to expand access to antiretroviral therapy (ART) and mental health services. However, efforts to implement task shared, SUD treatment and ART adherence interventions that can be feasibly and sustainably integrated into primary care are limited. Therefore, the purpose of this study is to help fill this gap in care by evaluating Khanya, a peer-delivered, behavioral intervention to improve HIV care outcomes and reduce substance use. The present study is a hybrid effectiveness-implementation trial designed to evaluate Khanya compared to usual care, enhanced with referral to a local outpatient substance use treatment program (Enhanced Standard of Care - ESOC) over 12 months. To provide care for those most in need, participants will be patients with HIV who are struggling with ART adherence and have elevated SUD risk. In this study, Khanya will be delivered as a stepped-care package in which the least resource-intensive part of the intervention (i.e., a single session problem solving intervention for HIV medication adherence) will be delivered first. Only individuals randomized to the Khanya intervention who are still struggling with HIV medication adherence after the first session will be stepped up to receive the more comprehensive, resource-intensive part of the intervention (i.e., six additional sessions of the intervention). Primary effectiveness outcomes in this clinical trial include ART adherence and SUD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive and on ART
* ≥18 years of age
* At least moderate substance use risk in the past 3 months for at least one non-tobacco substance (measured by the WHO- ASSIST: score ≥11 for alcohol, ≥4 for non-tobacco drugs)
* ART nonadherence and/or risk of virologic failure, defined as at least one of the following in the past 12 months 1) re-engaging in care after ≥1 month of being out of care (confirmed by pharmacy refill data) 2) ≥1 episodes of VL >400 copies/mL 3) on second- or third-line ARTs.

Exclusion Criteria:

* Severe risk/likely dependence for opiates (WHO ASSIST score >26) because opiate substitution therapy is largely not available
* Severe alcohol dependence symptoms that may warrant medical management of potential withdrawal symptoms/stabilization prior to study participation
* Inability to provide informed consent or complete study procedures in isiXhosa or English
* In third trimester of pregnancy during baseline
* Currently enrolled in another study or treatment program focused on substance use (including Matrix) or ART adherence.
* Untreated or undertreated major mental illness that would interfere with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in HIV Medication Adherence | Assessed from baseline through 12-month assessment
  Percentage of prescribed antiretroviral therapy (medications) taken as measured by real time wireless monitoring device (Wisepill)
Biological Measure of Substance Use | Assessed from baseline across 3-, 6-, and 12-month assessments
  Biomarker-verified substance use

SECONDARY OUTCOMES:
Changes in Self-Reported Substance Use | Assessed from baseline across 3-, 6-, and 12-month assessments
  Self-reported substance use will be assessed primarily by the World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (WHO-ASSIST). It is a measure used to assess substance use risk for alcohol, cannabis, cocaine, opiates, and amphetamines, hallucinogens, and other drugs. Standardized cutoff scores are used to categorize risk levels: low risk (0-3 for illicit drugs/0-10 for alcohol), moderate risk (4-26 for illicit drugs/11-26 for alcohol), or high risk (> 26) for substance use-related problems.
Biological Measure of Adherence | Assessed from baseline across 3-, 6-, and 12-month assessments
  Biomarker-confirmed ART adherence will be measured with Dried Blood Spot (DBS) testing
HIV Clinic Attendance | Assessed from baseline across 3-, 6-, and 12-month assessments
  Number of days participants in each condition were on-time to, late to, or missed an HIV clinic appointment (extracted from clinic records).
HIV Viral Load | Assessed from baseline across 6-, and 12-month assessments
  Percentage of patients with a detectable viral load
Employment Status Questionnaire | Assessed from baseline across 3-, 6-, and 12-month assessments
  Employment status of the participant with a range of locally appropriate response options including, but not limited to: working full-time, working part-time, unemployed or laid off and looking for work, in school or training, retired, disabled, in the military.

OTHER OUTCOMES:
Acceptability using a quantitative assessment based on RE-AIM | 3-month assessment
  15-item acceptability subscale of a pragmatic, quantitative assessment based on RE-AIM developed by the Applied Mental Health Research group (AMHR) at Johns Hopkins University. Total scores are averaged across all items and range from 0 to 3. Higher scores indicate greater acceptability.
Feasibility using a quantitative assessment based on RE-AIM | 3-month assessment
  16-item feasibility subscale of a pragmatic, quantitative assessment based on RE-AIM developed by the Applied Mental Health Research group (AMHR) at Johns Hopkins University. Total scores are averaged across all items and range from 0 to 3. Higher scores indicate greater acceptability.
Implementation Fidelity | From baseline over 6-months
  Independent fidelity ratings of a randomly selected subset (20%) of intervention sessions using a fidelity assessment developed for each session that includes 15-19 items that map onto each core intervention component, and factors unique to the peer delivery implementation strategy (i.e., appropriate self-disclosure, stigmatizing behaviors, common factors including warmth and non-judgment).
Uptake | From baseline over 6-months
  Uptake will be measured as an implementation outcome, including the % of patients who initiate treatment and treatment attendance.
Health-Related Quality of Life assessed by EQ-5D | Assessed from baseline across 3-, 6-, and 12-month assessments
  Health-related quality of life (HRQoL) will be measured with the EQ-5D which is the most widely used of the major HRQoL instruments capable of generating a single health utility index value to calculate quality-adjusted life-years (QALYs), and one of the most sensitive to changes in pain, physical and mental health functioning. This instrument measures HRQoL across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
CD4 Count | Assessed from baseline across 6-, and 12-month assessments
  Absolute CD4 value in the blood to measure immune function and disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, MS, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be uploaded to an NIH-supported data repository and available by request with appropriate permissions from PI.